CLINICAL TRIAL: NCT04867434
Title: A Double Blind, Randomized, Three Arm, Placebo-Controlled Phase 2b Study to Evaluate the Efficacy and Safety of RZL-012 in Subjects Seeking for Submental Fat Reduction
Brief Title: Efficacy and Safety of RZL-012 on Submental Fat Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raziel Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RZL-012-SMF-P2b-US-001
Record Dates: First submitted 2021-04-19; First posted 2021-04-30 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2021-04

CONDITIONS: Submental Fat
MeSH Terms: interventions — RZL-012

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RZL-012 50mg/ml (Active Comparator): Subjects treated with RZL-012 will undergo a single treatment session with 32±4 injections. The maximal number of injections will be 36 with maximal doses 270 mg for the high doses. Each injection point will be dosed with 7.5 mg for the high dose in a volume of 0.15 mL/injection site.
  Interventions: Drug: RZL-012
- RZL-012 34mg/ml (Active Comparator): Subjects treated with RZL-012 will undergo a single treatment session with 32±4 injections. The maximal number of injections will be 36 with maximal doses of 183.6 mg for the low dose. Each injection point will be dosed with 5.1 mg RZL-012 for the low dose in a volume of 0.15 mL/injection site.
  Interventions: Drug: RZL-012
- Placebo (Placebo Comparator): Placebo (vehicle) subjects will be injected with a 0.15 mL vehicle per each injection site. The maximal injection volume for all groups will be up to 5.4 mL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RZL-012 — small synthetic molecule for submental fat reduction
  Arms: RZL-012 34mg/ml; RZL-012 50mg/ml
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A total of 135 eligible male or female subjects will be randomized according to a predetermined randomization scheme (1:1:1 ratio) to receive a single multi-injection treatment of high dose RZL-012, low dose RZL-012, or placebo on Day 0. They will be monitored for safety and efficacy over 84 days.

DETAILED DESCRIPTION:
Each subject will be randomized to either active treatment (high or low dose RZL-012) or placebo at a ratio of 1:1:1 per group and receive one of the following:

* low dose (concentration of injected solution 34 mg/mL RZL-012) of 5.1 mg/0.15 mL/injection point that results in a dose/volume of 163.2±20.4 mg/4.8±0.6 mL RZL-012,
* high dose (concentration of injected solution 50 mg/mL RZL-012) of 7.5 mg/0.15 mL/injection point that results in a maximum total dose/volume of 240±30 mg/4.8±0.6 mL RZL-012,
* placebo of 0.15 mL/injection point that results in a total maximum volume of 4.8±0.6 mL.

Subjects treated with RZL-012 will undergo a single treatment session with 32±4 injections. The maximal number of injections will be 36 with maximal doses of 183.6 mg and 270 mg for the low and high doses, respectively. Each injection point will be dosed with 5.1 mg RZL-012 for the low dose or 7.5 mg for the high dose in a volume of 0.15 mL/injection site. Placebo (vehicle) subjects will be injected with a 0.15 mL vehicle per each injection site. The maximal injection volume for all groups will be up to 5.4 mL.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female subject between the ages of 18 and 65 years, inclusive.
2. Has body mass index (BMI) between >22 and <40.
3. Has SMF area that is contiguous and fits to 32±4 injections sites according to a grid with 1 cm distance between injection points.
4. Has moderate to severe grade 3 to 4 of SMF as rated by the C-SFS.
5. Has moderate to severe grade 3 to 4 of SMF as rated by the P-SFS.
6. Has stable weight, with no fluctuation of >5 kg in the past 12 months.
7. If female, is not pregnant or breastfeeding based on the following:

   * agree to the use of highly effective contraceptive methods for at least 2 weeks before baseline until 7 days after the last day of study drug and a negative serum pregnancy test (ß-hCG) at screening and negative urine pregnancy test at baseline; or
   * is of nonchildbearing potential defined as clinically infertile as the result of surgical sterilization (hysterectomy, bilateral tubal ligation, and/or bilateral oophorectomy); or
   * is confirmed postmenopausal status (defined as either having amenorrhea for ≥ 12 consecutive months without another cause and documented serum follicle-stimulating hormone (FSH) level > 40 mIU/mL or another documented medical condition (e.g., was born without a uterus)) NOTE: The following are considered highly effective contraceptive methods: hormonal oral contraceptives, injectables, and patches; intrauterine devices; double-barrier methods (synthetic condom, diaphragm, or cervical cap used with spermicidal foam, cream, or gel); and male partner sterilization.
8. If male (with or without vasectomy), agree to the use of highly effective contraceptive methods (as listed in Criterion #7 above) from study check-in until 7 days after the last day of study drug.
9. Is willing to avoid strenuous exercise for seven (7) days post treatment.
10. Is able to adhere to the visit schedule and protocol requirements and be available to complete the study.
11. Is willing and able to sign an Institutional Review Board (IRB) approved informed consent form (ICF) indicating that they are aware of the investigational nature of the study.

Exclusion Criteria:

Subjects must NOT meet any of the following Exclusion criteria to be eligible for enrollment:

1. Is unable to tolerate subcutaneous injections.
2. Has dysfunctional gallbladder activity (e.g., underwent cholecystectomy or cholecystitis).
3. Has any uncontrolled systemic disease that is not stabilized (i.e., cardiovascular disease, mental illness).
4. Has had treatment with botulinum toxin injections in the neck or chin area within nine (9) months prior to screening.
5. Has used anticoagulation therapies that may increase bleeding or bruising (i.e., aspirin, ibuprofen, vitamins, and herbal preparations) for seven (7) days prior to treatment.
6. Has skin laxity (i.e., elastosis, skin crepiness, skin redundancy, skin draping, vertical and/or horizontal skin bands and folds, blunting of cervical mental angle, loss of opposition of skin to underlying neck structures due to skin laxity) that could obscure the evaluation and treatment of SMF.
7. Has an extreme fat bulge under the chin and the submental fat was previously rated as 'very severe'.
8. Has fat extends down the neck beyond the Adam's Apple, towards the base of the neck where the fat extends laterally along the jawline making the jawline indistinguishable from the neck.
9. Has any scars, unshaven hair, tattoos, facial hair or jewelry on or near the proposed treatment area.
10. Has presence of structures or confounding factors that may interfere with assessing SMF such as but not limited to enlarged submandibular salivary and/or parotid glands, micrognanthia, chin implant, soft tissue volume augmentation of chin and/or jawline, pronounced platysmal bands and deep necklace lines or presence of facial jowls that could obscure the evaluation of SMF.
11. Has significant history or current evidence of a medical, psychological or other disorder that, in the Investigator's opinion, would preclude enrollment in the study.
12. Has an active dermatitis or open wound in the proposed treatment area.
13. Has abnormal coagulation tests (PT, PTT)
14. Has D-dimer value >0.64mg/L in screening visit
15. Has an active bacterial, fungal, or viral infection in the proposed treatment area.
16. Has a pre-existing skin condition in the submental region that, at the Investigator's discretion, may confound evaluation or analysis.
17. Has previously had treatments or surgery in the submentum, such as but not limited to, focused ultrasound, radiofrequency, cryolipolysis, liposuction, sodium deoxycholate, or neck lift.
18. Has pre-existing neurological or gastrointestinal condition leading to dysphagia, dysphonia, or facial nerve palsy.
19. Has Dercum's Disease
20. Has any pre-existing medical condition other than increased SMF that, at the Investigator's discretion, may result in increased submental fullness, such as but not limited to, thyroid enlargement, goiter, cervical lymphadenopathy, etc.
21. Has a planned fat reduction procedure of any variety to the submental region for the duration of the study.
22. Has medication or a history of coagulopathy.
23. Has a history or family history of venous thrombotic disease.
24. Has been treated chronically at least three (3) months prior to study entry with systemic steroids or immunosuppressive drugs.
25. Has been treated chronically at least one (1) week prior to study entry with non-steroidal anti-inflammatory drugs (NSAIDs).
26. Current participation or participation within three (3) months prior to the start of this study in a drug or other investigational research study.
27. Has claustrophobia or an MRI incompatible device or implant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raceli Gueta, PhD, Study Director — Raziel Therapeutics
Locations (1):
- DenovaResearch, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RZL-012 50mg/ml | RZL-012 34mg/ml | Placebo
Started | 50 | 53 | 48
Completed | 50 | 49 | 47
Not Completed | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RZL-012 50mg/ml | RZL-012 34mg/ml | Placebo | Total
Number analyzed (Participants) | 50 | 53 | 48 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (9.7) | 42.8 (10.7) | 41.6 (10.8) | 43 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 34 | 121
  Male | 8 | 8 | 14 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black Or African American | 5 | 4 | 5 | 14
  Race: White | 37 | 39 | 36 | 112
  Race: Asian | 4 | 5 | 5 | 14
  Race: American Indian Or Alaska Native | 1 | 3 | 1 | 5
  Race: Native Hawaiian Or Other Pacific | 0 | 1 | 1 | 2
  Race: Not reported or Unknown | 3 | 1 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 53 | 48 | 151

OUTCOME MEASURES:

1. Primary Outcome: Efficacy -Proportion of Subjects With at Least a 1-grade Improvement in the C-CAT Scale at Day 84
Description: To determine the efficacy of RZL-012 versus placebo on submental fat (SMF) reduction measured on Day 84 versus baseline using the Clinician Chin Assessment Tool (C-CAT). The CAT is composed of 5 points where 0 represents no fat and 4 represent very noticeable bulge and fat that extends beyond the neck
Time Frame: 84 days
Population: The proportion of subjects who have at least a 1-grade improvement in the C-CAT on Day 84 versus baseline will be calculated for the placebo group and the RZL-012 high-dose group along with 95% Confidence interval for proportion
Measure: Number; unit: participants
Arm/Group | RZL-012 50mg/ml | RZL-012 34mg/ml | Placebo
Number analyzed (Participants) | 50 | 53 | 48
participants | 43 | 39 | 27

2. Secondary Outcome: Efficacy - the Proportion of Subjects With at Least 1-grade Improvement in Subject Chin Assessment Tool (S-CAT)
Description: To determine the efficacy of RZL-012 versus placebo on submental fat (SMF) reduction measured on Day 84 versus baseline using the Subject Chin Assessment Tool (S-CAT). The CAT is composed of 5 points where 0 represents no fat and 4 represent very noticeable bulge and fat that extends beyond the neck
Time Frame: 84 days
Population: - The Chi-Square test will be applied to test the statistical difference between the placebo group and each of the RZL-012 dose groups in the responder rate at Day 84 where responder rate is defined as the percentage of subject achieving at least a 1-grade improvement from baseline in S-CAT
Measure: Number; unit: participants
Arm/Group | RZL-012 50mg/ml | RZL-012 34mg/ml | Placebo
Number analyzed (Participants) | 50 | 53 | 48
participants | 43 | 42 | 30

3. Secondary Outcome: Efficacy - Relative Change in Submental Fat Volume on Day 84 vs. Baseline
Description: Percent reduction from baseline in submental fat volume , as measured with MRI in RZL-012 treated subjects vs. placebo treated subjects on Day 84 following injection vs. baseline.
Time Frame: 84 days
Population: The Paired T-test for two means (paired observations) will be applied for testing the statistical significance of the change and percentage of change from baseline at Day 84 in SMF thickness measured with caliper and in SMF volume by MRI within each study group
Measure: Mean (Standard Deviation); unit: percentage of volume reduction
Arm/Group | RZL-012 50mg/ml | RZL-012 34mg/ml | Placebo
Number analyzed (Participants) | 41 | 44 | 45
percentage of volume reduction | -14.92 (9.98) | -8.34 (11.72) | 1.45 (8.68)

4. Secondary Outcome: Safety - Adverse Events Follow up
Description: To evaluate the safety of RZL-012 subcutaneous injections in the submental area, relative to placebo, as assessed by spontaneous adverse event reports and post injection evaluation of treatment area. Treatment area evaluations including, but not limited to evaluation of edema, bruising, dysphasia, dysphonia, erythema, dyspigmentation, induration, numbness, pain, paresthesia, and pruritus. The number of subjects with treatment-related adverse events will be compared within each treatment group, as assessed by CTCAE v4.0.
Time Frame: 84 days
Population: The incidence of AEs will be presented by treatment. Descriptive statistics will be calculated for quantitative data and frequency counts and percentages will be provided for categorical data. All reported AEs are treatment related
Measure: Number; unit: participants
Arm/Group | RZL-012 50mg/ml | RZL-012 34mg/ml | Placebo
Number analyzed (Participants) | 50 | 53 | 48
participants
  Dysphagia | 15 | 21 | 2
  Injection site edema | 21 | 27 | 27
  Injection site bruising | 18 | 17 | 20
  Injection site erythema | 7 | 4 | 3
  Injection site hemorrhage | 6 | 10 | 7
  Injection site hypoesthesia | 15 | 15 | 12
  Injection site mass | 5 | 4 | 1
  Injection site pain | 34 | 31 | 23
  Injection site paresthesia | 0 | 2 | 1
  Injection site pruritus | 5 | 5 | 6
  Injection site swelling | 17 | 18 | 16
  Localized edema | 10 | 6 | 3
  Injection site hypersensitivity | 2 | 1 | 0
  Injection site induration | 7 | 7 | 0
  Injection site movement impairement | 3 | 1 | 0
  Dizziness | 2 | 2 | 0
  Headache | 3 | 4 | 3
  Facial paralysis | 3 | 1 | 0
  Hypoesthesia | 3 | 0 | 0
  Dysphonia | 2 | 2 | 0
  Dyspnea | 2 | 2 | 0
  Induration | 1 | 1 | 1
  Injection site dermatitis | 0 | 0 | 1
  Injection site discomfort | 2 | 3 | 1
  Tenderness | 0 | 0 | 1
  Injection site nodule | 2 | 1 | 0
  Injection site warmth | 0 | 1 | 0
  pain | 4 | 4 | 0
  Swelling | 1 | 0 | 0
  Burning sensation | 0 | 0 | 1
  Facial nerve disorder | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: No difference from clinicaltrials.gov
Arm/Group | RZL-012 50mg/ml | RZL-012 34mg/ml | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/53 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/53 | 0/48
Other Adverse Events (participants affected / at risk) | 49/50 | 51/53 | 48/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RZL-012 50mg/ml (N=50) | RZL-012 34mg/ml (N=53) | Placebo (N=48)
Injection site edema (General disorders) | 21 | 27 | 27
Dysphagia (Gastrointestinal disorders) | 15 | 21 | 2
Injection site Bruising (General disorders) | 18 | 17 | 20
Injection site erythema (General disorders) | 7 | 4 | 3
Injection site hemorrhage (General disorders) | 6 | 10 | 7
Injection site hypoesthesia (General disorders) | 15 | 15 | 12
Injection site mass (General disorders) | 5 | 4 | 1
Injection site pain (General disorders) | 34 | 31 | 23
Injection site paraesthesia (General disorders) | 0 | 2 | 1
Injection site pruritus (General disorders) | 5 | 5 | 6
Injection site swelling (General disorders) | 17 | 18 | 16
Localized edema (General disorders) | 10 | 6 | 3
Injection site hypersensitivity (General disorders) | 2 | 1 | 0
Injection site induration (General disorders) | 7 | 7 | 0
injection site movement impairment (General disorders) | 3 | 1 | 0
dizziness (Nervous system disorders) | 2 | 2 | 0
headache (Nervous system disorders) | 3 | 4 | 3
facial paralysis (Nervous system disorders) | 3 | 1 | 0
hypoaesthesia (Nervous system disorders) | 3 | 0 | 0
dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
induration (General disorders) | 1 | 1 | 1
Injection site dermatitis (General disorders) | 0 | 0 | 1
Injection site discomfort (General disorders) | 2 | 3 | 1
Tenderness (General disorders) | 0 | 0 | 1
Injection site nodule (General disorders) | 2 | 1 | 0
Injection site warmth (General disorders) | 0 | 1 | 0
pain (General disorders) | 4 | 4 | 0
Swelling (General disorders) | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT04867434/Prot_001.pdf
  • Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT04867434/SAP_002.pdf